CLINICAL TRIAL: NCT01473914
Title: Trace Element Replenishment Study in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marcello Tonelli (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor-Investigator, Marcello Tonelli, MD, Professor, University of Alberta
Organization: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRSV1
Record Dates: First submitted 2011-09-23; First posted 2011-11-17 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Selenium; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose (Experimental): Standard renal vitamin plus low dose zinc and selenium plus vitamin E
  1 capsule p.o, daily
  Interventions: Dietary Supplement: Low dose: supplemental zinc, selenium and vitamin E; Dietary Supplement: Standard renal vitamin: B and C renal vitamin
- Medium dose (Experimental): Standard renal vitamin plus medium doses of zinc and selenium plus vitamin E
  1 capsule p.o, daily
  Interventions: Dietary Supplement: Standard renal vitamin: B and C renal vitamin; Dietary Supplement: Medium dose: supplemental zinc, selenium and vitamin E
- Standard treatment (Active Comparator): Standard renal vitamin
  1 capsule p.o, daily
  Interventions: Dietary Supplement: Standard renal vitamin: B and C renal vitamin

INTERVENTIONS:
Dietary Supplement: Low dose: supplemental zinc, selenium and vitamin E — 1. ZINC 25mg (AS ZINC SULFATE)
  2. SELENIUM 50 mcg (AS SODIUM SELENITE)
  3. VITAMIN E (D-ALPHA-TOCOPHEROL) (AS SUCCINATE) 250 IU
  Arms: Low dose
Dietary Supplement: Standard renal vitamin: B and C renal vitamin — 1. BIOTIN 300 MCG
  2. D-PANTOTHENIC ACID (CALCIUM D-PANTOTHENATE) 10 MG
  3. FOLIC ACID 1 MG
  4. NIACINAMIDE 20 MG
  5. VITAMIN B1 (THIAMINE MONONITRATE) 1.5 MG
  6. VITAMIN B12(CYANOCOBALAMIN) 6 MCG
  7. VITAMIN B2 (RIBOFLAVIN) 1.7 MG
  8. VITAMIN B6 (PYRIDOXINE HYDROCHLORIDE) 10 MG
  9. VITAMIN C (ASCORBIC ACID) 100 MG
  10. INERT FILLER (CORNSTARCH)
  Other Names: Replavite
Dietary Supplement: Medium dose: supplemental zinc, selenium and vitamin E — 1. ZINC 50 mg (AS ZINC SULFATE)
  2. SELENIUM 75 mcg (AS SODIUM SELENITE)
  3. VITAMIN E (D-ALPHA-TOCOPHEROL) (AS SUCCINATE) 250 IU
  Arms: Medium dose

SUMMARY:
A pilot randomized trial that compares a new renal nutritional supplement with the standard renal vitamin.

The primary objective is to compare two doses (medium and high) of the new supplement with the renal vitamin currently being prescribed to people with End Stage Renal Disease (ESRD).

Secondary objective is to demonstrate the feasibility of recruitment for a definitive larger trial.

DETAILED DESCRIPTION:
People with severe kidney disease follow a restricted diet aimed at reducing intake of sodium, potassium and phosphate. These dietary restrictions require reducing their intake of many fresh fruits and vegetables, which may lead to nutritional deficiency. Although the potential for malnutrition in people with kidney disease is well recognized, blood levels of most vitamins and trace elements are rarely measured. Instead, most North Americans with severe kidney disease are routinely prescribed a "renal vitamin" such as Replavite which contains a mixture of B and C vitamins.

Recent evidence (including our work; see http://www.biomedcentral.com/bmcmed/subjects/nephrology) indicates that people with severe kidney disease are often deficient in several other biologically essential substances (selenium, zinc) that are readily amenable to supplementation. Pilot data from the Northern Alberta Renal Program (NARP) indicate that approximately 90% of patients have zinc levels below the lower limit of normal; findings for selenium are similar.

Potential benefits of zinc supplementation include improvements in immune function, taste sensitivity (perhaps reducing dietary sodium intake), and improved appetite. Potential benefits of selenium supplementation include reductions in the risk of vascular disease and infection. Supplementation with vitamin E was shown in a randomized trial to reduce serious cardiovascular morbidity in people with kidney failure, but is not routinely used in dialysis patients. This suggests that supplementation of zinc, selenium, and vitamin E has theoretical benefits in kidney failure. Since patients with kidney failure already take many medications, it is logical to combine any new nutritional supplements with the ingredients of the standard renal vitamin to reduce pill burden.

This protocol concerns a novel nutritional supplement consisting of zinc, selenium and vitamin E in addition to the contents of the standard renal supplement of B and C vitamins.

This pilot randomized, double blind trial will compare 2 doses of the new supplement with the standard renal vitamin.

2.0 Objectives: Primary objective: compare two formulations of the new supplement (low and medium doses of zinc and selenium) with standard treatment (Replavite or equivalent renal vitamin).

Secondary objective: demonstrate the feasibility of recruitment for a definitive larger trial

ELIGIBILITY:
Inclusion Criteria:

1. Stable on hemodialysis for 3 to 36 months
2. Age greater or equal to 18 years
3. Receiving Replavite or equivalent renal vitamin at baseline
4. Receiving 3 dialysis treatments per week

Exclusion Criteria:

1. Pregnant (sexually active pre-menopausal females must have negative serum pregnancy test at baseline)
2. Pregnancy, kidney transplantation, a dialysis modality switch, or gastrointestinal surgery planned within 6 months
3. Known allergy to corn starch
4. Known allergy to zinc, selenium, vitamin E or renal vitamin.
5. Projected life expectancy of <6 months
6. Any other conditions or procedures that, in the opinion of the investigator, would impede absorption of the study product.
7. Participants already taking a vitamin E, zinc or selenium supplement (alone or included in another multi-vitamin).
8. Individuals with a history of head or neck cancer in the past 5 years.
9. Ostomy or short gut syndrome.
10. Enroll in another (interventional) trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with zinc deficiency | 90 days following baseline
  Proportion of participants with zinc deficiency in the combined experimental arms compared to the proportion of participants with zinc deficiency in the active comparator arm.

SECONDARY OUTCOMES:
Proportion of participants with zinc deficiency | 180 days following baseline
  The proportion of participants with zinc deficiency in each arm compared to each other arm at each time point.
Proportion of participants with selenium deficiency | 90 days and 180 days following baseline
  The proportion of participants with selenium deficiency in each arm compared to each other arm at each time point.
Zinc | 90 days and 180 days following baseline
  Zinc concentration in each arm compared to each other arm.
Selenium | 90 days and 180 days following baseline
  Selenium concentration measured in each arm compared to each other arm.

OTHER OUTCOMES:
Proportions of participants with serious adverse events | 30 days following last day of intervention
  The proportion of participants in each arm compared to each other arm experiencing serious adverse events resulting in death, life threatening illness, hospitalization or prolongation of existing hospitalization, or persistent or significant disability.
Proportion of participants with adverse events | 30 days following last day of intervention
  The proportion of participants with adverse events (and by each type of adverse event) in each arm compared to each other arm.
Change in interdialytic weight | 90 days and 180 days following baseline
  Change in interdialytic weight in each arm compared to each other arm.
Salt sensitivity | 90 days and 180 days following baseline
  The proportion of participants with recognized and detect salt sensitivities in each arm compared to each other arm.

CONTACTS AND LOCATIONS:
Overall Officials: Marcello A Tonelli, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tonelli M, Wiebe N, Thompson S, Kinniburgh D, Klarenbach SW, Walsh M, Bello AK, Faruque L, Field C, Manns BJ, Hemmelgarn BR; Alberta Kidney Disease Network. Trace element supplementation in hemodialysis patients: a randomized controlled trial. BMC Nephrol. 2015 Apr 11;16:52. doi: 10.1186/s12882-015-0042-4. PMID 25884981
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- See also: Published open access article with final results — http://bmcnephrol.biomedcentral.com/articles/10.1186/s12882-015-0042-4